CLINICAL TRIAL: NCT07260747
Title: Comparison of the Effects of Virtual Reality-Based Interventions on Foot Function, Foot Pressure, and Balance in Sedentary Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-78097791-020-4737
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Foot Diseases
Keywords: exercise; foot
MeSH Terms: conditions — Foot Diseases; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR Biodex Group (Experimental): This group will participate in a virtual reality-supported rehabilitation program integrated with the Biodex Balance System device. Participants will perform interactive balance and postural stability exercises through this system
  Interventions: Other: VR Biodex Group
- Video-Based VR Group (Active Comparator): Participants in this group will perform balance and foot exercises accompanied by exercise videos containing visual guidance. This intervention aims to provide the virtual reality experience through video-based content.
  Interventions: Other: Video-Based VR Group
- Control Group (Active Comparator): This group will follow a traditional home exercise program without any virtual reality intervention. This group will serve as a baseline for comparing the results of the other two groups
  Interventions: Other: Control Group

INTERVENTIONS:
Other: VR Biodex Group — This group will participate in a virtual reality-supported rehabilitation program integrated with the Biodex Balance System device.
  Arms: VR Biodex Group
Other: Video-Based VR Group — : Participants in this group will perform balance and foot exercises accompanied by exercise videos containing visual guidance.
  Arms: Video-Based VR Group
Other: Control Group — This group will follow a traditional home exercise program without any virtual reality intervention.
  Arms: Control Group

SUMMARY:
Comparison of the Effects of Virtual Reality-Based Interventions on Foot Function, Foot Pressure, and Balance in Sedentary Individuals

ELIGIBILITY:
Inclusion Criteria:

* Sedentary Individual
* Individuals between the ages of 18-25
* Being a university student

Exclusion Criteria:

* Athletes
* Individuals with orthopedic or neurological problems.
* Surgery history
* Cognitive impairment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Foot Function Assessment | 6 weeks
  Foot pain, disability, and activity limitation will be assessed using the Foot Function Index (FFI), a validated 23-item questionnaire. The total FFI score ranges from 0 to 100, with higher scores indicating worse foot function (greater pain, disability, and activity limitation).
Foot Pressure Assessment - Maximum Plantar Pressure | 6 weeks
  Plantar pressure during standing and walking will be assessed using a pedobarographic measurement system. Maximum plantar pressure will be recorded, with higher values indicating greater localized loading on the foot.
Foot Pressure Assessment - Contact Area | 6 weeks
  The pedobarographic system will measure the total plantar contact area during standing and walking. Larger contact area values indicate greater surface area participation in load distribution.
Foot Pressure Assessment - Center of Pressure (COP) | 6 weeks
  The pedobarographic system will measure center of pressure displacement during standing and walking. COP path characteristics provide objective indicators of stability and gait mechanics; greater displacement typically indicates reduced postural control.
Balance Performance Assessment | 6 weeks
  Static and dynamic balance performance will be assessed using the Biodex Balance System. The system provides balance scores ranging from 0 to 12, where lower scores indicate better balance performance.
Physical Activity Level Assessment | 6 weeks
  Physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ) - Short Form. Weekly metabolic equivalent of task (MET-minutes/week) will be calculated to classify physical activity as low, moderate, or high. Higher MET-minutes/week indicate higher physical activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceşehir University Health Center, Istanbul, Turkey (Türkiye)